CLINICAL TRIAL: NCT04048083
Title: Effect of Mental and Computer-aided Training of Reaching and Grasping Movements on Motor Control Processes in People With Bilateral Upper Limb Congenital Transverse Deficiency
Brief Title: Computer-aided and Mental Trainings Induced Plasticity of Sensorimotor Cortex in Patients Born Without Upper Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Wrocław University of Science and Technology (Other); Kessler Foundation (Other); Nencki Institute of Experimental Biology, Warsaw, Poland (Unknown); Hospital of St. Hedwig in Trzebnica (Unknown)
Responsible Party: Principal Investigator, Jaroslaw Marusiak, Co-Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DEC-2011/03/B/NZ7/00588
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Amelia of Upper Limb
Keywords: bilateral upper limb congenital transverse deficiency; neuroplasticity; sensorimotor cortex; mental training; virtual environment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients-MT (Experimental): 3 Patients with bilateral upper limb congenital transverse deficiency that participated in kinesthetic mental training (MT) of reaching to grasp movements
  Interventions: Behavioral: Mental trainings
- Patients-CAT (Experimental): 3 Patients with bilateral upper limb congenital transverse deficiency that participated in computer-aided training (CAT) of reaching to grasp movements using virtual environment with visual-feedback.
  Interventions: Behavioral: Computer-aided trainings
- Patients-CAMT (Experimental): 3 Patients with bilateral upper limb congenital transverse deficiency that participated in kinesthetic mental training of reaching to grasp movements supplemented by virtual environment (patients that received both types of training).
  Interventions: Behavioral: Computer-aided and mental trainings
- Healthy-controls (Active Comparator): 9 Healthy, age and gender-matched subjects, without any kind of training
  Interventions: Other: No trainings

INTERVENTIONS:
Behavioral: Mental trainings — Patients will receive 36 trainings (12 weeks with 3 trainings a week) of mental, kinesthetic reaching-to-grasp movement. During each training session they will perform 3 practice trials by following the instructions, after practicing 3 trials, the instructions will be discontinued, and subjects will perform 30 mental movements by following auditory cues.
  Arms: Patients-MT
Behavioral: Computer-aided trainings — Patients will receive 36 trainings (12 weeks with 3 trainings a week) of visual feedback of reaching-to-grasp movement. During each training session they will be sitting on a chair, in front of a computer screen observing simple tasks of reaching and precision fine grasping of a small object with 4 fingers of virtual upper extremity using the visualization software that will be coded specifically for the purpose of this experiment.
  Arms: Patients-CAT
Behavioral: Computer-aided and mental trainings — Patients will receive 36 trainings (12 weeks with 3 trainings a week) of mental, kinesthetic reaching-to-grasp movement that will be supplemented by visual feedback of this task by the visualization software that will be coded specifically for the purpose of this experiment (they will receive trainings that link the features of the two mentioned above types of training (MT and CAT).
  Arms: Patients-CAMT
Other: No trainings — Healthy controls without any kind of training
  Arms: Healthy-controls

SUMMARY:
This project will explore a potentially powerful trainings that may be administered before upper extremity transplantation to induced plasticity of sensorimotor cortex in humans with congenital absence of upper limbs. We believe that engaging this population to computer-aided and/or mental trainings would facilitate structural and functional reorganization of the brain to promote motor function recovery.

DETAILED DESCRIPTION:
This project will explore a potentially powerful trainings that may be administered before upper extremity transplantation to induced plasticity of sensorimotor cortex in humans with congenital absence of upper limbs.

Our aim is to compare neurophysiological outcome of bilateral upper limb congenital transverse deficiency humans who are engaged in different types of training (mental-MT, computer-aided training-CAT and subjects receiving both type of trainings-CAMT). We hypothesize that all forms of training provide plastic changes in sensorimotor cortex. Specifically, we hypothesize that for CAMT group we will observe more prompt CNS-reorganization as compared to MT and CAT groups.

Our second aim is to examine mechanisms of neural and muscular system plasticity underlying neurophysiological function reorganization following the specific training and also to develop a computer system for training subjects through visual biofeedback. The control procedure of virtual upper extremity should be realized through recognition of intention of hand motion based on biosignals analysis.

Our protocol contains twelve weeks of trainings with three training sessions during a week (on Monday, Wednesday and Friday) and four measurement sessions (before the training period - PRE, after 4 weeks of trainings - POST4, after 8 weeks of trainings - POST8 and after 12 weeks of training - POST12).

Based on different methods we will use, we would like to ewaluate: structural changes in CNS, functional changes in CNS, functional changes in peripheral nervous system and functional changes in muscles of upper extremity stump by comparing results to the pre-training (PRE) values (with results from POST4, POST8 and POST12) and across the groups.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age between 18 and 25 years
* Health status: bilateral upper limb congenital transverse deficiency individuals. Subjects must be free from neurological impairment. The subjects must have no current or past history of central or peripheral nervous system dysfunction, be taking no current medication known to affect the neuromuscular system, have no greater than moderate consumption of alcohol or caffeine, and be able to remain seated for 1 hour 30 min and lay supine without moving for 30 min (MRI test). All recruited subjects will be interviewed and their health status and medical history will be evaluated by a medical practitioner qualified to practice surgery and transplant surgery.
* Training history: Subjects not participating in any type of training program in the last 5 years
* Right Hemispheric Dominance. We will use Foot Dominance test - Observation of our subjects to see which foot they use to kick a ball, step up onto a stair, and step onto a coin placed on the floor.
* Availability and interest: All candidates for the study must be available for the familiarization, training, and testing sessions and must have transportation to these sessions.

Exclusion Criteria for patients:

* Presence of neurological impairment (history of central or peripheral nervous system dysfunction)
* Taking medication that affects the neuromuscular system
* Left hemispheric dominance
* Participation in training over the last five years

Inclusion Criteria for control subjects:

* Age between 18 and 25 years
* Health status: subjects must be free from neurological and neuromuscular system impairment. The subjects must have no current or past history of central or peripheral nervous system dysfunction, be taking no current medication known to affect the neuromuscular system, have no greater than moderate consumption of alcohol or caffeine, and be able to remain seated for 1 hour 30 min and lay supine without moving for 30 min (MRI test). ). All recruited subjects will be interviewed and their health status and medical history evaluated by neurologist.
* Training history: subjects not participating in any type of training program in the last 5 years.
* Hemispheric Dominance -right. We will use The Edinburgh inventory (Oldfield, 1971) and Foot Dominance test.
* Availability and interest - All subjects for the study must be available for the familiarization, training, and testing sessions and must have transportation to these sessions.

Exclusion Criteria for control subjects:

* Presence of neurological impairment (history of central or peripheral nervous system dysfunction)
* Taking medication that affects the neuromuscular system
* Left hemispheric dominance
* Participation in training over the last five years

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-03-11 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Before trainings period (PRE)
  To evaluate structural changes in central nervous system (CNS) the MRI method will be used
Magnetic Resonance Imaging (MRI) | After 4 weeks of trainings period (POST4)
  To evaluate structural changes in central nervous system (CNS) the MRI method will be used
Magnetic Resonance Imaging (MRI) | After 8 weeks of trainings period (POST8)
  To evaluate structural changes in central nervous system (CNS) the MRI method will be used
Magnetic Resonance Imaging (MRI) | After 12 weeks of trainings period (POST12)
  To evaluate structural changes in central nervous system (CNS) the MRI method will be used
Functional Magnetic Resonance Imaging (fMRI) | Before trainings period (PRE)
  To evaluate functional changes in CNS, the fMRI will be used
Functional Magnetic Resonance Imaging (fMRI) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in CNS, the fMRI will be used
Functional Magnetic Resonance Imaging (fMRI) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in CNS, the fMRI will be used
Functional Magnetic Resonance Imaging (fMRI) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in CNS, the fMRI will be used
Transcranial magnetic stimulation (TMS) | Before trainings period (PRE)
  To evaluate excitability of the sensory-motor cortex of the brain.
Transcranial magnetic stimulation (TMS) | After 4 weeks of trainings period (POST4)
  To evaluate excitability of the sensory-motor cortex of the brain.
Transcranial magnetic stimulation (TMS) | After 8 weeks of trainings period (POST8)
  To evaluate excitability of the sensory-motor cortex of the brain.
Transcranial magnetic stimulation (TMS) | After 12 weeks of trainings period (POST12)
  To evaluate excitability of the sensory-motor cortex of the brain.
Electroencephalography (EEG) | Before trainings period (PRE)
  To evaluate functional changes in CNS, the 128-channels EEG will be used.
Electroencephalography (EEG) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in CNS, the 128-channels EEG will be used.
Electroencephalography (EEG) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in CNS, the 128-channels EEG will be used.
Electroencephalography (EEG) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in CNS, the 128-channels EEG will be used.
Near-infrared spectroscopy (NIRS) | Before trainings period (PRE)
  To evaluate functional changes in peripheral nervous system.
Near-infrared spectroscopy (NIRS) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in peripheral nervous system.
Near-infrared spectroscopy (NIRS) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in peripheral nervous system.
Near-infrared spectroscopy (NIRS) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in peripheral nervous system.
Electromyography (EMG) | Before trainings period (PRE)
  To evaluate functional changes in muscles of upper extremity stump
Electromyography (EMG) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in muscles of upper extremity stump
Electromyography (EMG) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in muscles of upper extremity stump
Electromyography (EMG) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in muscles of upper extremity stump
Mechanomyography (MMG) | Before trainings period (PRE)
  To evaluate functional changes in muscles of upper extremity stump
Mechanomyography (MMG) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in muscles of upper extremity stump
Mechanomyography (MMG) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in muscles of upper extremity stump
Mechanomyography (MMG) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in muscles of upper extremity stump
Temperature measurements (Temp) | Before trainings period (PRE)
  To evaluate functional changes in muscles of upper extremity stump
Temperature measurements (Temp) | After 4 weeks of trainings period (POST4)
  To evaluate functional changes in muscles of upper extremity stump
Temperature measurements (Temp) | After 8 weeks of trainings period (POST8)
  To evaluate functional changes in muscles of upper extremity stump
Temperature measurements (Temp) | After 12 weeks of trainings period (POST12)
  To evaluate functional changes in muscles of upper extremity stump

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kisiel-Sajewicz, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences
Locations (1):
- University School of Physical Education in Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurzynski M, Jaskolska A, Marusiak J, Wolczowski A, Bierut P, Szumowski L, Witkowski J, Kisiel-Sajewicz K. Computer-aided training sensorimotor cortex functions in humans before the upper limb transplantation using virtual reality and sensory feedback. Comput Biol Med. 2017 Aug 1;87:311-321. doi: 10.1016/j.compbiomed.2017.06.010. Epub 2017 Jun 15. PMID 28641235
- [Derived] Mencel J, Marusiak J, Jaskolska A, Kaminski L, Kurzynski M, Wolczowski A, Jaskolski A, Kisiel-Sajewicz K. Motor imagery training of goal-directed reaching in relation to imagery of reaching and grasping in healthy people. Sci Rep. 2022 Nov 3;12(1):18610. doi: 10.1038/s41598-022-21890-1. PMID 36329083
- [Derived] Mencel J, Jaskolska A, Marusiak J, Kaminski L, Kurzynski M, Wolczowski A, Jaskolski A, Kisiel-Sajewicz K. Motor Imagery Training of Reaching-to-Grasp Movement Supplemented by a Virtual Environment in an Individual With Congenital Bilateral Transverse Upper-Limb Deficiency. Front Psychol. 2021 Mar 22;12:638780. doi: 10.3389/fpsyg.2021.638780. eCollection 2021. PMID 33828507